CLINICAL TRIAL: NCT02601066
Title: Identification of Predictors of Cardiac Arrhythmias and Sudden Death in Pediatric Patients Affected With Laminopathies
Brief Title: Cardiac Arrhythmias and Sudden Death in Patients Affected With Laminopathies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Sant Joan de Deu (Other)
Collaborators: Marcio Andres Foundation (Other)
Responsible Party: Principal Investigator, Georgia Sarquella Brugada, MD PhD, MD, PhD, Hospital Sant Joan de Deu
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CARDIO-2015-01 LMNA
Record Dates: First submitted 2015-10-26; First posted 2015-11-10 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Cardiomyopathy Associated With Myopathy and Sudden Death
Keywords: LMNA; Sudden Death; Neuromuscular
MeSH Terms: conditions — Cardiomyopathy Associated With Myopathy And Sudden Death; Death, Sudden

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EPS and ECG holter monitor (Experimental): Electrophysiological study (EPS) and ECG holter monitor implantation
  Interventions: Device: Electrophysiological Study and ECG holter monitor

INTERVENTIONS:
Device: Electrophysiological Study and ECG holter monitor — Electrophysiological Study and ECG holter monitor implantation

SUMMARY:
This research study includes patients ages 1 to 25 years old with Lamin A/C related muscular dystrophy (LMNA-MD). The goal of this study is to evaluate how the heart is affected in children and teens with LMNA-MD. The evaluation includes an echocardiogram, an electrocardiogram, an electrophysiological study and the implantation of a subcutaneous ECG holter monitor.

DETAILED DESCRIPTION:
The LMNA related muscular dystrophies are monogenic progressive neuromuscular disorders. Affected pediatric patients can present at birth or in childhood and are classified as either congenital muscular dystrophy (LMNA-CMD), congenital onset Limb-girdle muscular dystrophy type 1B (LGMD1B) or childhood onset Emery Dreifuss muscular dystrophy (EDMD). These distinct clinical presentations all involve variants in the LMNA gene and can be distinguished by method of inheritance. Those with LMNA-CMD have new mutations in the LMNA gene not carried by either parent, while those with LGMD1B and EDMD will have a parent who may or not have symptoms with the same variant (change in the LMNA gene). There is no current cure or treatment for LMNA-MD.

While heart involvement has been studied for the adult forms of LMNA muscular dystrophy. These studies have identified an increased risk for arrhythmia (abnormal heart rhythms), conduction defects, cardiomyopathy and sudden cardiac death. To date there has been no study evaluating the age of onset of heart involvement, the type of heart involvement, the rate of heart disease progression and the risk of sudden cardiac death in children affected with LMNA-MD. The investigators' research aims to evaluate heart involvement in children and teens affected by LMNA-MD.

This is a prospective interventional natural history study. The intervention consists of 3 steps: 1) High complexity echocardiography, 2) Electrophysiological Study, 3) subcutaneous ECG holter monitor implantation.

The duration of the active protocol will last 3 years. Potential subjects will be identified through the Spanish muscular dystrophy network and the Congenital Muscle Disease International Registry. The study will involve one on-site visit at Sant Joan de Déu Hospital in Barcelona, Spain; and a yearly follow-up that will be arrange individually (either a second visit to Barcelona or doctors will travel to see the patient).

At Visit 1, subjects will have their baseline assessments, including an echocardiogram, an electrocardiogram, a electrophysiological study and medication review and the subcutaneous ECG holter monitor implantation.

The second study visit will occur 12-14 months after the first study visit. Remote monitoring through the holter device will continue for 36 months after placement of the device.

For those individuals traveling from outside Spain, travel arrangements will be eased by Andres Marcio Foundation

ELIGIBILITY:
Inclusion Criteria:

* Age of onset of muscle weakness between birth and 5 years of age
* Confirmed LMNA related muscular dystrophy by gene mutation AND clinical history

Exclusion Criteria:

* ny neuromuscular disorder other than LMNA related muscular dystrophy
* unable to comply with an echocardiogram or an electrophysiologic study

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-12 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Ejection Fraction (%) | 4 years
  Heart involvement has been studies for the adult forms of LMNA muscular dystrophy. These studies have identified an increased risk for arrhythmia (abnormal heart rhythms), conduction defects, cardiomyopathy and sudden cardiac death. To date there has been no study evaluating the age of onset of heart involvement, the type of heart involvement, the rate of heart disease progression and the risk of sudden cardiac death in children affected with LMNA-MD.
  Outcome Measures: Ejection Fraction%, Strain Rate, time of arrhythmia in 24 hours, type of arrhythmia.
Strain (%) | 4 years
  Myocardial deformation (strain) can be obtained based on Tissue Doppler Imaging (TDI) or on bidimensional images (speckle tracking). TDI allows better time definition and can be also used in case of poor echocardiographic windows. Analyses from bidimensional images allow assessment of radial and circumferencial strain, as well as apical and basal rotation, needed to calculate ventricular torsion. Normal values of longitudinal LV deformation are between -20 to -25 %.
Strain Rate (%/s) | 4 years
  Rate of myocardial deformation in time. Diastolic myocardial deformation can be assessed more clearly in this way. Normal values of longitudinal LV deformation are 1 - 1.5/s or higher.
Presence of arrhythmias (yes/no) | 3 years
  By inserting the Holter monitoring system, presence or absence of arrhythmias can be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Sarquella-Brugada, MD, PhD, Principal Investigator — Hospital Sant Joan de Deu
Locations (1):
- Pediatric Arrhythmia Unit, Hospital Sant Joan de Déu, Esplugues, Barcelona, Spain